CLINICAL TRIAL: NCT03757208
Title: Effect of Preoperative Oral Carbohydrate Loading on Recovery in Patients Undergoing Day-case Cholecystectomy. A Randomised Controlled Trial.
Brief Title: Preoperative Carbohydrate Loading in Patients Undergoing Day-case Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Heli Helminen, Principal Investigator, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uoulu 192/2012
Record Dates: First submitted 2018-11-20; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Preoperative Care
Keywords: Carbohydrate loading, oral carbohydrate beverage

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (No Intervention)
- Carbohydrate rich drink (CHD) group (Active Comparator)
  Interventions: Dietary Supplement: carbohydrate rich drink

INTERVENTIONS:
Dietary Supplement: carbohydrate rich drink — The carbohydrate rich drink (CHD) group received oral carbohydrate (200 ml) 2-3 h before surgery,
  Arms: Carbohydrate rich drink (CHD) group

SUMMARY:
Background: Preoperative carbohydrate loading has been shown to reduce preoperative discomfort and postoperative nausea and vomiting in general surgical patients. Few studies have been focused on patients undergoing day-case surgery.

Objective: The aim of this prospective randomized study was to determine whether preoperative carbohydrate loading enhanced the recovery of patients undergoing day-case cholecystectomy.

Design: A randomised controlled trial. Setting: Secondary care in a district general and a university hospital in Finland between 2013-2016.

Patients: A total of 113 patients ASA physical status I or II (18-70 yr) undergoing day-case cholecystectomy were included in the study. Exclusion criteria were bleeding or coagulation disorders, BMI >40, dementia, insulin-treated diabetes, migraine, Meniere's disease or a history of alcohol or drug abuse.

Intervention: The carbohydrate rich drink (CHD) group received oral carbohydrate (200 ml) 2-3 h before surgery, and the control (Fasting) group fasted from midnight according to standard protocol.

Main outcome measures: Visual analogue scales (VAS) were used to score six discomfort parameters. The needs for analgesia or antiemetics, the time to drinking, eating and first mobilization after surgery, and the time to discharge and hospital readmission were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 yr (ASA physical status I-II) eligible for day-case cholecystectomy

Exclusion Criteria:

* Patients with bleeding or coagulation disorders, BMI >40, dementia or suffering from insulin-treated diabetes, migraine, Meniere's disease or with history of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-04-08 (Actual); Primary Completion 2016-05-16 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Number of given pain and antiemetic medication (n) | One day (in recovery room after operation to discharge time)
Thirst, hunger, dryness of mouth, tiredness, nausea, and pain (Visual analogue scale, VAS 0-100) | One day (4 hours after operation and at discharge)
Time of drinking, eating and first mobilisation (minutes after operation) | One day (in recovery room after operation to discharge time)
Time of discharge (hours after operation) | One day (time of discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Haukipuro, Ph.M.D, Study Chair — University Hospital of Oulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Helminen H, Branders H, Ohtonen P, Saarnio J. Effect of pre-operative oral carbohydrate loading on recovery after day-case cholecystectomy: A randomised controlled trial. Eur J Anaesthesiol. 2019 Aug;36(8):605-611. doi: 10.1097/EJA.0000000000001002. PMID 31021880